CLINICAL TRIAL: NCT03512886
Title: The Effect of Multiple-Task Training on Physical and Cognitive Functions in Patients With Multiple Sclerosis
Brief Title: The Effect of Multiple-Task Training in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Cagla Ozkul, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 231
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Multi-task training; Balance; Mobility; Cognition; Upper extremity function
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single task training (Active Comparator): The exercise program consisting of 10 different motor tasks will be implemented in a single task training group.
  Interventions: Other: Single task training
- Multi-task training (Experimental): In the multitasking training group, a second motor task in the first two weeks, a cognitive task in the third and fourth week, both motor and cognitive tasks in the last two weeks will be added to these 10 different motor tasks.
  Interventions: Other: Multi-task training
- Control group (No Intervention): The control group will be taught relaxation exercises and will be asked to perform the exercises at home.

INTERVENTIONS:
Other: Multi-task training — In the multitasking training group, a second motor task in the first two weeks, a cognitive task in the third and fourth week, both motor and cognitive tasks in the last two weeks will be added to these 10 different motor tasks.
  Arms: Multi-task training
Other: Single task training — An exercise program consisting of 10 different motor tasks will be implemented in a single task training group.
  Arms: Single task training

SUMMARY:
The Activities of Daily Living requires the ability to perform multiple activities at the same time, not just the motor or cognitive activity. When many tasks are performed at the same time, the attention capacity is effectively used and attention is shared according to the difficulty and priority of the tasks. There is evidence that patients with Multiple Sclerosis (MS) have reduced performance during multitasking.

In this study, the investigators aim to investigate the effect of multitasking training on balance, mobility, upper extremity performance and cognitive functions in patients with MS.

DETAILED DESCRIPTION:
Patients with MS between 0-1,5 score according to the Extended Disability Status Scale (EDSS) will be included in the study. The balance, mobility, upper extremity performance, the cognitive function will be evaluated twice.

The study was designed as a prospective, randomized controlled study. The patients will be randomly assigned to three groups, the "multi-task training (MT)" group, the "single task training (ST)" group, and "control" group. The training will be twice a week for 6 weeks.

Statistical analyses will be performed using the SPSS software version 15 (SPSS Inc. Chicago, IL, USA). The pre-training and post-training measurements of groups will be compared with the Wilcoxon Test. The significance level was set at p< 0.05

ELIGIBILITY:
Inclusion Criteria:

* Participants who are ambulatory and volunteer to participate to the study, in a stable phase of the disease, without relapses in the last 3 month, with an EDSS between 0-1,5.

Exclusion Criteria:

* Participants who have orthopedic, vision, hearing, or perception problems

  * Patients who have any cardiovascular or pulmonary disease in which exercise is contraindicated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Mobility | ten minutes]
  Timed Up and Go Test
Modified Sensory Organization Test | Fifteen minutes]
  The Modified Sensory Organization Test, which is performed using computerized posturography, measures postural sway in response to 4 different sensory conditions is measured using a force platform.
Upper extremity function | ten minutes
  9-Hole Peg Test
cognitive function | thirty minutes
  The Brief Repeatable Battery of Neuropsychological Tests

SECONDARY OUTCOMES:
Physical Activity | ten minutes
  International Physical Activity Questionnaire- Long version
Fatigue Impact | five minutes
  Fatigue impact scale consists of forty questions and evaluates the effects of fatigue on the 3 dimensions of daily life activities; cognitive function, physical function and psychosocial function. Each question is graded between 0 (no problem) and 4 (maximum problem).
Fatigue Severity | Five minutes
  In the Fatigue Severity Scale (FSS), participants are asked to rate their fatigue level between 1 and 7 in the 9 statements (including motivation, exercise, physical functioning, carrying out duties, and interfering with work, family, or social life) during the last week.
Balance Confidence | five minutes
  Activities-specific Balance Confidence (ABC) is a scale in which the patient rates his perceived level of confidence while performing 16 daily living activities.
Neuropsychological Questionnaire | one minute
  Multiple Sclerosis Neuropsychological Questionnaire - MSNQ

CONTACTS AND LOCATIONS:
Overall Officials: Cagla Ozkul, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silsupadol P, Siu KC, Shumway-Cook A, Woollacott MH. Training of balance under single- and dual-task conditions in older adults with balance impairment. Phys Ther. 2006 Feb;86(2):269-81. PMID 16445340
- [Background] Pashler H. Dual-task interference in simple tasks: data and theory. Psychol Bull. 1994 Sep;116(2):220-44. doi: 10.1037/0033-2909.116.2.220. PMID 7972591
- [Background] Tombu M, Jolicoeur P. A central capacity sharing model of dual-task performance. J Exp Psychol Hum Percept Perform. 2003 Feb;29(1):3-18. doi: 10.1037//0096-1523.29.1.3. PMID 12669744
- [Background] Wajda DA, Sosnoff JJ. Cognitive-motor interference in multiple sclerosis: a systematic review of evidence, correlates, and consequences. Biomed Res Int. 2015;2015:720856. doi: 10.1155/2015/720856. Epub 2015 Mar 9. PMID 25839039
- [Background] Sosnoff JJ, Wajda DA, Sandroff BM, Roeing KL, Sung J, Motl RW. Dual task training in persons with Multiple Sclerosis: a feasability randomized controlled trial. Clin Rehabil. 2017 Oct;31(10):1322-1331. doi: 10.1177/0269215517698028. Epub 2017 Mar 20. PMID 28933609
- [Background] Hofheinz M, Mibs M. The Prognostic Validity of the Timed Up and Go Test With a Dual Task for Predicting the Risk of Falls in the Elderly. Gerontol Geriatr Med. 2016 Mar 16;2:2333721416637798. doi: 10.1177/2333721416637798. eCollection 2016 Jan-Dec. PMID 28138492
- [Background] Oxford Grice K, Vogel KA, Le V, Mitchell A, Muniz S, Vollmer MA. Adult norms for a commercially available Nine Hole Peg Test for finger dexterity. Am J Occup Ther. 2003 Sep-Oct;57(5):570-3. doi: 10.5014/ajot.57.5.570. PMID 14527120
- [Background] Boringa JB, Lazeron RH, Reuling IE, Ader HJ, Pfennings L, Lindeboom J, de Sonneville LM, Kalkers NF, Polman CH. The brief repeatable battery of neuropsychological tests: normative values allow application in multiple sclerosis clinical practice. Mult Scler. 2001 Aug;7(4):263-7. doi: 10.1177/135245850100700409. PMID 11548987
- [Background] Benedict RH, Munschauer F, Linn R, Miller C, Murphy E, Foley F, Jacobs L. Screening for multiple sclerosis cognitive impairment using a self-administered 15-item questionnaire. Mult Scler. 2003 Feb;9(1):95-101. doi: 10.1191/1352458503ms861oa. PMID 12617275
- [Background] Armutlu K, Korkmaz NC, Keser I, Sumbuloglu V, Akbiyik DI, Guney Z, Karabudak R. The validity and reliability of the Fatigue Severity Scale in Turkish multiple sclerosis patients. Int J Rehabil Res. 2007 Mar;30(1):81-5. doi: 10.1097/MRR.0b013e3280146ec4. PMID 17293726
- [Background] Armutlu K, Keser I, Korkmaz N, Akbiyik DI, Sumbuloglu V, Guney Z, Karabudak R. Psychometric study of Turkish version of Fatigue Impact Scale in multiple sclerosis patients. J Neurol Sci. 2007 Apr 15;255(1-2):64-8. doi: 10.1016/j.jns.2007.01.073. Epub 2007 Mar 6. PMID 17337007
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Derived] Ozkul C, Eldemir K, Apaydin Y, Gulsen C, Irkec C, Guclu-Gunduz A. Effects of multi-task training on motor and cognitive performances in multiple sclerosis patients without clinical disability: a single-blinded randomized controlled trial. Acta Neurol Belg. 2023 Aug;123(4):1301-1312. doi: 10.1007/s13760-023-02172-7. Epub 2023 Jan 7. PMID 36609834